CLINICAL TRIAL: NCT06003803
Title: Effects of Self-Regulated Digital Learning on Competence in Motivational Interviewing on Patients' Medication Adherence Among Psychiatric Mental Health Nurses
Brief Title: Digital Learning on Competence in Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen I Liu, Distinguished Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: digital learning
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-12

CONDITIONS: Nurse's Role; Motivation
Keywords: digital learning; motivational interviewing; self-regulation
MeSH Terms: conditions — Self-Control | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- digital learning in motivational interviewing (Experimental): Receive digital learning in motivational interviewing for three months, once a week, 40 minutes each time
  Interventions: Behavioral: digital learning in motivational interviewing
- conventional education (No Intervention): Receive conventional education for three months.

INTERVENTIONS:
Behavioral: digital learning in motivational interviewing — Receive digital learning in motivational interviewing for three months, once a week, 40 minutes each time
  Arms: digital learning in motivational interviewing

SUMMARY:
Motivational interviewing is an essential practical skill to promote medication adherence; however, it is rarely emphasised in nursing education. Purposes: 1. To develop a self-regulated digital learning system for motivational interviewing; 2. To evaluate the effectiveness of digital learning of motivational interviewing on mental health nurses' knowledge, skills and self-efficacy (confidence); 3. To compare the effectiveness of self-regulated digital learning, blended learning and treatment as usual learning.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric registered nurse

Exclusion Criteria:

* nursing administrator
* expected to resign within three months
* blended learners who have participated in motivational interviewing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
motivational interviewing skill | The time point of measurement is the baseline, the change in the 3month after the intervention, and the change in the 6 month]
  Motivational Interviewing skill is a 12-items assessment tool.Total scores is range between 0 and 12, with a higher score indicating better skill.

SECONDARY OUTCOMES:
Motivational Interviewing Knowledge and Attitudes Test (MIKAT) | The time point of measurement is the baseline, the change in the 3month after the intervention, and the change in the 6 month]
  Motivational Interviewing Knowledge and Attitudes Test is a 29-items self-reporting scales.Total scores on the MIKAT range between 0 and 29, with a higher score indicating better knowledge.
Motivational Interviewing Confidence Survey (MICS) | The time point of measurement is the baseline, the change in the 3month after the intervention, and the change in the 6 month]
  MICS is a 24-items self-reporting with 10-point Likert scale.Total scores on the MICS range between 0 and 240, with a higher score indicating better self-efficacy.

OTHER OUTCOMES:
self-regulation scale for Taiwanese college students (TSSRQ) | The time point of measurement is the baseline, the change in the 3month after the intervention, and the change in the 6 month]
  TSSRQ is a 39-items self-reporting with a higher score indicating better self-regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan